CLINICAL TRIAL: NCT05333406
Title: Open-label, Dose-escalation, Phase 1 Clinical Trial to Determine the Safety and Dose of EN001 in Patients With Charcot-Marie-Tooth Disease (CMT) Type 1A
Brief Title: Determine the Safety and Dose of EN001 in Patients With Charcot-Marie-Tooth Disease (CMT) Type 1A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ENCell (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENCell_2020_02
Record Dates: First submitted 2022-01-06; First posted 2022-04-19 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Charcot-Marie-Tooth Disease, Type IA
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose group A (Low dose) (Experimental): Participants will receive EN001 intravenously (IV) once on Day 0.
  Interventions: Drug: EN001
- Dose group B (High dose) (Experimental): Participants will receive EN001 intravenously (IV) once on Day 0.
  Interventions: Drug: EN001

INTERVENTIONS:
Drug: EN001 — EN001 intravenously (IV) in the treatment of Charcot-Marie-Tooth disease (CMT) type 1A Dosage for each group is as follows.
  Dose group A (Low dose): 5.0x10^5 cells/kg
  Other Names: EN001 (allogeneic umbilical cord-derived mesenchymal stem cells)
  Arms: Dose group A (Low dose)
Drug: EN001 — EN001 intravenously (IV) in the treatment of Charcot-Marie-Tooth disease (CMT) type 1A Dosage for each group is as follows.
  Dose group B (High dose): 2.5x10^6 cells/kg
  Other Names: EN001 (allogeneic umbilical cord-derived mesenchymal stem cells)
  Arms: Dose group B (High dose)

SUMMARY:
Open-label, Dose-escalation, Phase 1 Clinical Trial to Determine the Safety and Dose of EN001 in Patients with Charcot-Marie-Tooth disease (CMT) type 1A

DETAILED DESCRIPTION:
It is the first in human (FIH), 3+3 design clinical trial to evaluate the safety and tolerability and determine the maximum tolerated dose (MTD) of EN001 (allogeneic umbilical cord-derived mesenchymal stem cells) in the treatment of Charcot-Marie-Tooth disease (CMT) type 1A.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 19 to 75 years old
2. Those diagnosed with CMT type 1A by a genetic test
3. Those whose CMTNS-v2 score is more than 2 and 20 or fewer points, and the severity of the disease is mild to moderate
4. Those who have dorsiflexion muscle weakness
5. Those who can comply with the requirements for clinical trials
6. For women of childbearing potential, those who have a negative urine pregnancy test at screening
7. Those who use a medically acceptable method of contraception until clinical trial visit 7 (short-term follow-up visit, 16 weeks): hormonal contraception, intrauterine device (IUD), intrauterine system (IUS), vasectomy, tubal ligation, or double barrier method using a cervical cap or a diaphragm with a male condom.
8. Those who voluntarily agree to participate in this study and sign an IRB-approved consent form after being informed about the characteristics of this clinical trial prior to all screening tests

Exclusion Criteria:

1. Those with other neuromuscular diseases that the investigator judges cannot participate in the clinical trial
2. Patients diagnosed with type 1 or type 2 diabetes
3. Those with a history of stroke or cerebral ischemic attack within 12 months of screening
4. Those with a history of coronary artery diseases such as myocardial infarction or unstable angina within 12 months of screening
5. Those who have undergone orthopedic surgery on the lower extremities (bone and ligament correction, artificial joint insertion, osteotomy, arthroscopic surgery) within 6 months of screening
6. Those who have ankle contractures or have surgery that may affect muscle strength assessment
7. Those who have experience with stem cell therapy or gene therapy before screening
8. Those who have participated in clinical trials for chemical synthetic drugs before screening (except when 5 times the half-life has passed)
9. Patients with uncontrolled hypertension (If the systolic blood pressure is 180 mmHg or higher or the diastolic blood pressure is 110 mmHg or higher)
10. If there is a history of malignant tumors other than basal cell carcinoma or squamous cell carcinoma occurring in the skin within 5 years of screening
11. Those who diagnosed with active pulmonary tuberculosis
12. Immunosuppressed patients who are taking immunosuppressants, chemotherapy, radiation therapy, etc.
13. Mental illness patients
14. Those who are pregnant or lactating
15. Those with significant heart, lung, liver, kidney, hematological, immunological, behavioral disease, or other clinically significant diseases including malignant tumors
16. Those who have a previous or current medical condition that may adversely affect the safety of the subject, make it difficult to complete treatment or affect the evaluation of clinical trial results at the discretion of the investigator
17. Those who do not have the will or ability to comply with clinical trial procedures at the discretion of the investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Number of participants of any Adverse Events (AEs)/Serious Adverse Events (SAEs) related investigational product | Week 16 after treatment
  Number of participants with treatment-related AEs/SAEs as assessed by CTCAE v5.0
Determination of Dose-limiting toxicity (DLT) levels of EN001 | Up to Week 4 after dosing on Day 0
  Among the adverse events occurring for 4 weeks after administration of the investigational product, Grade 3 or higher adverse events according to CTCAE v5.0
Determination of Maximum tolerated dose (MTD) levels of EN001 | Up to Week 4 after dosing on Day 0
  Among the adverse events occurring for 4 weeks after administration of the investigational product, Grade 3 or higher adverse events according to CTCAE v5.0 Maximum tolerated dose defines the evaluated maximum dose level in which greater than two participants of six participants experience Dose-limiting toxicity (DLT) under the dose level. The dose level where two participants of six participants experience DLT will be the maximum tolerated dose.
Number of participants with Vital Signs abnormalities | From screening up to Week 16
  Vital Signs include blood pressure (mmHg), pulse (times/minute), respiratory rate (times/minute), and body temperature (℃) and will be assessed by CTCAE v 5.0 to evaluate safety and tolerability of EN001.
  The number of participants with at least one potentially clinically significant abnormal vital sign finding were reported as treatment emergent adverse events (TEAEs).
Number of participants with clinically significant abnormalities of Physical Examinations | From screening up to Week 16
  Physical Examinations include general appearance, head, ears/eyes/nose/throat, cardiovascular, respiratory, abdomen, skin, lymph nodes, extremities, musculoskeletal and neurologic and will be assessed by CTCAE v 5.0 to evaluate safety and tolerability of EN001.
  Number of participants with potentially clinically significant abnormalities in physical examinations were reported as TEAEs.
Number of participants with abnormalities of Laboratory Parameters | From screening up to Week 16
  Laboratory Parameters include hematology, chemistry laboratory tests, urinalysis, coagulation test and plasma viral load test and will be assessed by CTCAE 5.0 to evaluate safety and tolerability of EN001.
  Number of participants with at least one potentially clinically significant abnormal finding were reported as TEAEs.
Number of participants with 12-lead Electrocardiography (ECG) abnormalities | From screening to baseline on Day 1 (Predose to end of infusion and 90 min after completion of infusion)
  Measured by result of the ECG measurements and findings

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | From screening to the end of treatment/withdrawal visit (up to approximately 5 years per subject)
  Occurrence of any adverse reactions, development of new blood clots, tumors, immune responses (like autoimmune reactions) and death, and/or serious adverse events related investigational product will be summarized by actual treatment groups respectively.
Number of participants with abnormalities of Vital Signs, Physical Findings, and Laboratory Parameters | From screening to the end of treatment/withdrawal visit (up to approximately 5 years per subject)
  Abnormalities of Vital Signs, Physical Findings, and Laboratory parameters (as described above) will be collected and analyzed, and then assessed by CTCAE 5.0 to evaluate the long-term safety of EN001.
Change from baseline in disease severity CMTNS-v2 score | Screening and baseline on Day 0 (up to approximately 5 years per subject after Week 4)
  Disease severity measured by CMTNS-v2 score will be collected and analyzed to evaluate the exploratory efficacy of EN001.
Change from baseline in gait and balance functions | Screening and baseline on Day 0 (up to approximately 5 years per subject after Week 4)
  Gait and balance functions measured by Ten Meter Walking Test(10MWT), Functional Disability Scale (FDS), and Overall Neuropathy Limitation Score (ONLS) leg scale will be collected and analyzed to evaluate the exploratory efficacy of EN001.
Change from baseline in the degree of muscle damage (%) | Screening and baseline on Day 0 (up to approximately 5 years per subject after Week 4)
  The degree of muscle damage measured by lower extremity magnetic resonance imaging (MRI) scan will be collected and analyzed to evaluate the exploratory efficacy of EN001.
Change from baseline in nerve regeneration potential | Screening and baseline on Day 0 (up to approximately 5 years per subject after Week 4)
  Nerve generation potential measured by MNCV, SNCV, CMAP, and SNAP will be collected and analyzed to evaluate the exploratory efficacy of EN001.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea